CLINICAL TRIAL: NCT06625515
Title: A Phase 1/2, Open-Label, Dose-Escalation and Expansion First-In-Human Study of ATX-559, an Oral Inhibitor of the Helicase DHX9, in Patients With Locally Advanced or Metastatic Solid Tumors and Molecularly Defined Cancers
Brief Title: First-in-Human Study of ATX-559, an Oral Inhibitor of DHX9, in Patients With Advanced or Metastatic Solid Tumors, and Molecularly Defined Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by sponsor based on the adverse event profile.
Sponsor: Accent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATX-559-001
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors; Breast Cancer Recurrent; Colorectal Cancer Metastatic; Colon Cancer; Rectal Adenocarcinoma; Endometrial Cancer
Keywords: MSI-high/dMMR tumors; BRCA1 mutation; BRCA2 mutation; DHX9; dMMR; deficient mismatch repair; microsatellite instability
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Endometrial Neoplasms; Microsatellite Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation (Experimental): Subjects will be enrolled at various doses or schedules of ATX-559 to identify the RP2D
  Interventions: Drug: ATX-559
- Dose Expansion: MSI-H/dMMR solid tumors (Experimental)
  Interventions: Drug: ATX-559
- Dose Expansion: BRCA1- or BRCA2-deficient HER2-negative breast cancer (Experimental)
  Interventions: Drug: ATX-559

INTERVENTIONS:
Drug: ATX-559 — DHX9 tablets will be taken orally

SUMMARY:
The goal of this study is to identify a safe and tolerated dose of the orally administered DHX9 inhibitor ATX-559. In addition, this study will evaluate the pharmacokinetics, pharmacodynamics and preliminary antitumor activity of ATX-559 in patients with advanced solid tumors and molecularly defined cancers.

DETAILED DESCRIPTION:
ATX-559 is an oral drug that inhibits a protein called DHX9, a multi-functional RNA helicase that is involved in the maintenance of genomic stability by resolving DNA/RNA secondary structures that may lead to DNA replication stress and DNA damage in certain molecularly defined cancers. ATX-559 has been shown preclinically to induce robust anti-tumor activity of a variety of different solid tumors, including models with BRCA deficiency and microsatellite instability-high (MSI-H) and/or deficient mismatch repair (dMMR).

This is a first-in-human, Phase 1, open-label, single-arm, dose-escalation and expansion study to:

Evaluate the safety profile of ATX-559 and determine the recommended phase 2 dose (RP2D). In addition, the study aims to characterize the PK, PD, and preliminary anti-tumor activity of orally administered ATX-559. Exploratory objectives include examination of biomarker responses in relationship to ATX-559 exposure.

Patients with molecularly selected locally advanced or metastatic solid tumors (for example, BRCA1- or BRCA2-deficient breast cancer and solid tumors with microsatellite instability (MSI-H) and/or deficient mismatch repair (dMMR) will be enrolled to preliminarily assess the anti-tumor effect, and further examine the safety and PK of ATX-559 at the RP2D.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with histologically confirmed solid tumors who have locally recurrent or metastatic disease
* Refractory to or relapsed after all standard therapies with proven clinical benefit, unless as deemed by the Investigator, the subject is not a candidate for standard treatment, there is no standard treatment, or the subject refuses standard treatment after expressing an understanding of all available therapies with proven clinical benefit
* For the expansion cohorts, participants must have histological confirmation of the specified tumor types:
* BRCA1 or BRCA2 deficient, HER2 negative metastatic breast cancer
* dMMR or MSI-H with unresectable or metastatic solid tumors
* There is no limit to the number of prior treatment regimens
* Have measurable or evaluable disease
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Key Exclusion Criteria:

* Clinically unstable central nervous system (CNS) tumors or brain metastasis
* Any other concurrent anti-cancer treatment
* Has undergone a major surgery within 3 weeks of starting study treatment
* Medical issue that limits oral ingestion or impairment of gastrointestinal function that is expected to significantly reduce the absorption of ATX-559
* Clinically significant (ie, active) or uncontrolled cardiovascular disease
* Unable to transition off strong or moderate CYP2C8 inhibitors or inducers
* Pregnancy or intent to breastfeed or conceive a child within the projected duration of treatment

Other inclusion and exclusion criteria as defined in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) of ATX-559 | 12 months
  Identification of a tolerable and safe dose for expansion cohorts based on dose limiting toxicities
Safety and tolerability of ATX-559 | 12 months
  Incidence of adverse events graded according to CTCAE v5.0

SECONDARY OUTCOMES:
Preliminary evidence of antitumor activity | 12 months
  Objective response rate based on RECIST v1.1
Pharmacodynamic activity of ATX-559 in blood over time via measurement of circBRIP1 RNA levels | 12 months
Maximum observed plasma concentration of ATX-559 (Cmax) | 12 months
Calculated time to reach maximum observed plasma concentration (Tmax) | 12 months
Calculated area under the plasma concentration-time curve of ATX-559 (AUC0-t) | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado Cancer Center - Anschutz Medical Campus,, Aurora, Colorado
  - Stephenson Cancer Center at OU Medicine, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No